CLINICAL TRIAL: NCT06395415
Title: Development of a Mobile Health Intervention for Electronic Cigarette Use Among Young Adults
Acronym: EQUIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB21-1839
Record Dates: First submitted 2024-04-26; First posted 2024-05-02 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Electronic Nicotine Delivery Systems; Tobacco Products; Cigarette Smoking
MeSH Terms: conditions — Vaping; Cigarette Smoking | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mobile health (mHealth) (Experimental): Participants in this arm will receive a 6-week mHealth message based intervention through their smartphone. They will also have the option of requesting free nicotine replacement therapy (NRT) throughout the treatment period.
  Interventions: Behavioral: EQUIP
- Standard care (Active Comparator): Participants in this arm will receive a 5-10 minute walk-through of electronic nicotine delivery system (ENDS) and tobacco education and skills based on the most recent evidence. They will also have the options of requesting a sample of NRT.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: EQUIP — The intervention is delivered directly to participants' mobile phones using the Insight® platform, which allows for the implementation of assessments and interventions. Insight has been used in prior mHealth studies and allows for the delivery of tailored content based on parameters, such as intervention stage. The intervention has two stages: 1) Motivational enhancement (weeks 1-2) and 2) Skills and information (weeks 3-6). The first stage of messages will utilize personalized feedback and motivational interviewing prompts, while the second stage will provide health information on ENDS and skills, such as deep breathing. Content is tailored to motivation level (low/medium or high) and dual use status.
  Arms: mobile health (mHealth)
Behavioral: Standard Care — Those in the standard advice group will be given offered a sample of NRT, instruction on its use, and will be encouraged to use in conjunction with standard web-based resources on ENDS and cessation over the course of a ten minute walk-through with study staff.
  Arms: Standard care

SUMMARY:
Electronic Nicotine Delivery Systems (ENDS) use remains prevalent among young adults, and many have high interest in quitting, yet research on effective intervention is lacking. A mobile health (mHealth) intervention that translates effective smoking cessation materials and pharmacotherapy may be a promising avenue for intervention. The initial phase of the proposed study uses a pilot study to evaluate a novel mHealth intervention for young adult ENDS and dual product (ENDS and combustible cigarette) users.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-26 years old, ability to understand the English language, willing and able to provide informed consent
2. Current ENDS user (at least 4 out of 7 days per week of use for the past one month); for focus groups, at least half of participants will report current cigarette smoking (at least 1 cigarette per day on at least 1 day per week in the past month)
3. Report interest in quitting or reducing ENDS (at least 6/10 scale in interest of quitting or reducing
4. Does not currently (in past one year) meet criteria for major psychiatric disorder including severe alcohol or substance use disorder (excluding tobacco use disorder), schizophrenia, bipolar disorder, and obsessive compulsive disorder
5. For women, not currently pregnant, planning to become pregnant, or breastfeeding due to lack of information on ENDS use and possible harms from NRT during pregnancy
6. Not currently using smoking cessation medication (i.e., Varenicline, Bupropion
7. No history of adverse reactions to nicotine replacement therapy

Exclusion Criteria:

1. Does not own a mobile phone or is unwilling to receive text messages to their device
2. No interest in quitting or reducing use of ENDS
3. Uses electronic cigarettes less than 4 days per week in the past month
4. Reports past-year serious psychiatric illness, including severe alcohol or substance use disorder (excluding tobacco use disorder), schizophrenia, bipolar disorder, and obsessive compulsive disorder
5. Is currently using smoking cessation medication including Varenicline or Bupropion
6. Are a female who is currently pregnant or nursing or planning to become pregnant within the next 6 months

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
ENDS cessation | post-treatment (6 weeks) and at 6-week follow-up (week 12).
  ENDS cessation will be measured using a modified Timeline Followback Interview using 7-day point prevalence abstinence with study staff and then confirmed via a mailed saliva cotinine test.

SECONDARY OUTCOMES:
ENDS use | post-treatment (6 weeks) and at 6-week follow-up (week 12).
  Frequency of ENDS use as determined by Timeline Followback Interview with study staff will be measured as a secondary outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago BREATHE Laboratory, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
Interested parties can contact the PI for access to deidentified participant data. Requests will be granted as appropriate.